CLINICAL TRIAL: NCT00985361
Title: Effect of Vitamin D Supplementation on Hemoglobin A1c in Patients With Uncontrolled Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ProMedica Health System (Other)
Responsible Party: Mate Soric, ProMedica
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09-055
Record Dates: First submitted 2009-09-25; First posted 2009-09-28 (Estimated); Last update posted 2010-05-06 (Estimated); Status verified 2009-10

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D 2000 international units daily (Experimental)
  Interventions: Dietary Supplement: Vitamin D3 2000 international units daily
- Vitamin C 500mg daily (Active Comparator)
  Interventions: Dietary Supplement: Vitamin C 500mg daily

INTERVENTIONS:
Dietary Supplement: Vitamin D3 2000 international units daily — Vitamin D3 2000 international unit tablets once daily for 3 months
  Arms: Vitamin D 2000 international units daily
Dietary Supplement: Vitamin C 500mg daily — Vitamin C 500mg tablets once daily for 3 months
  Arms: Vitamin C 500mg daily

SUMMARY:
The purpose of this study is to determine if daily supplementation with 2000 International Units of Vitamin D will improve hemoglobin A1c in uncontrolled type 2 diabetics.

DETAILED DESCRIPTION:
Vitamin D is typically understood to support musculoskeletal health when administered concomitantly with calcium. A number of recent studies suggest, however, that this important nutrient may play a significant role in many pathophysiological processes, including diabetes mellitus. With the prevalence of diabetes mellitus ever increasing, novel mechanisms for controlling blood glucose and hemoglobin A1c are being sought to help prevent the costly and debilitating complications of this chronic disease.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Hemoglobin A1c >7% measured in the 3 months prior to randomization
* Age 21 to 75 years

Exclusion Criteria:

* Renal insufficiency (defined as CrCl <30mL/min)
* Gestational diabetes
* Malabsorption syndrome
* Patients taking vitamin D supplements at doses >400 international units daily

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2009-10; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Mate M Soric, PharmD, Principal Investigator — ProMedica Health System
Locations (3):
- United States (3):
  - Flower Hospital Family Medicine Residency, Sylvania, Ohio
  - Center for Health Services, Toledo, Ohio
  - Toledo Hospital Family Medicine Residency, Toledo, Ohio

REFERENCES:
- [Derived] Soric MM, Renner ET, Smith SR. Effect of daily vitamin D supplementation on HbA1c in patients with uncontrolled type 2 diabetes mellitus: a pilot study. J Diabetes. 2012 Mar;4(1):104-5. doi: 10.1111/j.1753-0407.2011.00164.x. No abstract available. PMID 22018074